CLINICAL TRIAL: NCT05914662
Title: Phase II Clinical Study of Zanubrutinib Combined With Bendamustine and Rituximab (ZBR) for Time-limited Treatment of Waldenstrom Macroglobulinemia
Brief Title: Zanubrutinib Plus BR in Newly Diagnosed Symptomatic WM
Acronym: ZBR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022070
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom macroglobulinemia; Zanubrutinib; newly diagnosed
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: Patients were treated with ZBR regimen for 6 cycles, followed by Zanubrutinib monotherapy for 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib, bendamustine, rituximab combination therapy Group (Experimental): Patients were treated with ZBR regimen for 6 cycles, followed by zanubrutinib monotherapy for an additional 6 months.
  Interventions: Drug: Zanubrutinib, Bendamustine and Rituximab

INTERVENTIONS:
Drug: Zanubrutinib, Bendamustine and Rituximab — Zanubrutinib, 160mg orally, twice a day; Bendamustine 70 mg/m2 on days 1 and 2 of each cycle; Rituximab (375 mg/m2 intravenously on day 0 of each cycle. ZBR was administered every 4 weeks for a total of 6 cycles, followed by maintenance therapy with zanubrutinib monotherapy for another 6 months.

SUMMARY:
This study aims to evaluate the long-term efficacy of BTK inhibitor Zanubrutinib combined bendamustine and rituximab (ZBR) for time-limited treatment of Waldenstrom macroglobulinemia, The combination therapy is expected to improve the remission depth, prolong the remission time, and improve the progression-free survival and overall survival of newly diagnosed WM patients. On the one hand, the patients have to bear a long-term economic burden, which is often difficult for some patients to adhere to for a long time. On the other hand, in the course of long-term treatment of BTKi, drug resistance and intolerable side effects are prone to occur. At the same time, it can prevent the disease rebound after the withdrawal of BTKi, so as to achieve the phased withdrawal of WM

DETAILED DESCRIPTION:
WM not only has the characteristics of lymphoma, such as lymphadenopathy, hepatosplenomegaly, and tumor cells expressing CD20, but also has the characteristics of myeloma, such as secreting monoclonal IgM, and tumor cells expressing plasma cell differentiation marker CD38, etc. Clinical studies have also shown that BR regimen and BTK inhibitor zanubrutinib are effective for WM.

This study aims to evaluate the long-term efficacy of BTK inhibitor Zanubrutinib combined bendamustine and rituximab (ZBR) for time-limited treatment of Waldenstrom macroglobulinemia, The combination therapy is expected to improve the remission depth, prolong the remission time, and improve the progression-free survival and overall survival of newly diagnosed WM patients. On the one hand, the patients have to bear a long-term economic burden, which is often difficult for some patients to adhere to for a long time. On the other hand, in the course of long-term treatment of BTKi, drug resistance and intolerable side effects are prone to occur. At the same time, it can prevent the disease rebound after the withdrawal of BTKi, so as to achieve the phased withdrawal of WM. This prospective phase II study was designed to evaluate the rate of deep response in newly diagnosed symptomatic WM. Eligible patients received ZBR for 6 cycles followed by zanubrutinib monotherapy for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The gender of the patient is not limited, and the age is ≥18 years old;
* Must meet WM's diagnostic standards;
* The patient is an untreated or patient who has not undergone standard treatment.
* The specific conditions are as follows:

  1. No combined chemotherapy with BTKi, BR, RCD, VRD, CHOP and COP
  2. No treatment regimen containing fludarabine
  3. Chlorambucil or cyclophosphamide for less than 4 weeks (alone or in combination with adrenal glucocorticoids)
  4. The above treatment did not reach the treatment response (MR)
  5. If the above treatment has been applied, the treatment needs to be stopped for 2 weeks before entering the group to start treatment
* The indications for the treatment of indolent lymphoma mainly include (at least one of the following conditions):

  1. Symptomatic hyperviscosity;
  2. Symptomatic peripheral neuropathy;
  3. Amyloidosis;
  4. Cold agglutinin disease; cryoglobulinemia;
  5. Disease-related cytopenia (Hb<100 g/L, PLT<100×10^9/L);
  6. Giant lymph nodes;
  7. Those with systemic systemic symptoms: for two weeks/recurrent fever (above 38℃) and not caused by infection, or Night sweats and/or weight loss >10% within 6 months;
  8. The disease progresses rapidly, for example, the lymph nodes increase by more than 50% within 2 months, and/or peripheral blood lymphocytes absolute value doubling time <6 months, and/or rapid hemoglobin or platelet non-autoimmune causes slow down
  9. When there is evidence that the disease has transformed.
* ECOG score ≤ 2 points
* Laboratory examination: neutrophils ≥ 0.75×10^9/L; platelets ≥ 50×10^9/L; total bilirubin ≤ 2.5 times upper limit; alanine aminotransferase/aspartate aminotransferase ≤3 times upper limit. Creatinine clearance rate ≥ 30ml/min.
* The patient's expected survival time is ≥ 3 months.

Exclusion Criteria:

* Malignant tumors (including active central nervous system lymphoma) other than B-NHL have been diagnosed or treated within the past year;
* There is clinical evidence that large cell lymphoma transformation has occurred;
* Non-lymphoma-related liver and kidney damage: alanine aminotransferase (ALT)> 3 times the upper limit of normal value, aspartate aminotransferase (AST)> 3 times the upper limit of normal value, total bilirubin (TBIL)> upper limit of normal value 2 Times, serum creatinine clearance rate <30ml/min;
* Other serious medical conditions will affect the study (such as uncontrolled diabetes, gastric ulcers, other serious cardiopulmonary diseases, etc.). The decision-making power belongs to the researcher;
* Known history of infection with human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics.
* Central nervous system dysfunction with clinical manifestations or central invasion (Bing-Neel syndrome);
* Patients who have undergone major surgery (not including lymph node biopsy) within the past 14 days or expected major surgery during treatment;
* Inability to swallow capsules or suffer from malabsorption syndrome, diseases that significantly affect gastrointestinal function, have undergone gastric or small bowel resection, symptomatic inflammatory bowel disease or ulcerative colitis, partial or complete intestinal obstruction.
* Need to receive strong cytochrome P450 (CYP) 3A inhibitor treatment.
* Women who are pregnant or breastfeeding, women of childbearing age who have not taken contraception;
* Allergy to the drugs used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Best combined complete response (CR) and very good partial response (VGPR) | up to the end of 12 cycles of treatment(each cycle is 28 days)
  To evaluate the efficacy of zanubrutinib plus bendamustine and rituximab (ZBR) regimen in the treatment of newly diagnosed WM patients, mainly the best deep response rate, namely the best deep response rate (VGPR and above).

SECONDARY OUTCOMES:
Overall objective response rate (ORR), complete response rate(CR),major response rate(MR) | up to the end of 12 cycles of treatment(each cycle is 28 days)
  using criteria from 6th international workshop on WM
Time to response, time to best response | up to the end of 12 cycles of treatment(each cycle is 28 days)
  Defined as after initiation of treatment， the time interval between the first documented remission of disease
Overall survival(OS) | Up to 3 years after the end of treatment
  3-year OS rate after treatment
Progression free survival(PFS) | Up to 3 years after the end of treatment
  3-year PFS rate after treatment
Duration of Response | Up to 3 years after the end of treatment
  DOR is defined as the time from the first occurrence of overall response (CR, PR or MR) until disease progression or death due to any cause.
Time to Next Treatment | Up to 3 years after the end of treatment
  Defined as the amount of time from the start of trial until the patient requires a new form of treatment to treat their WM
Safety of treatment regimens | Up to 3 years after the end of treatment
  Defined as Treatment-related adverse reactions in patients receiving treatment under this study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739
- [Background] Dimopoulos MA, Garcia-Sanz R, Gavriatopoulou M, Morel P, Kyrtsonis MC, Michalis E, Kartasis Z, Leleu X, Palladini G, Tedeschi A, Gika D, Merlini G, Kastritis E, Sonneveld P. Primary therapy of Waldenstrom macroglobulinemia (WM) with weekly bortezomib, low-dose dexamethasone, and rituximab (BDR): long-term results of a phase 2 study of the European Myeloma Network (EMN). Blood. 2013 Nov 7;122(19):3276-82. doi: 10.1182/blood-2013-05-503862. Epub 2013 Sep 4. PMID 24004667
- [Background] Castillo JJ, Meid K, Gustine JN, Leventoff C, White T, Flynn CA, Sarosiek S, Demos MG, Guerrera ML, Kofides A, Liu X, Munshi M, Tsakmaklis N, Xu L, Yang G, Branagan AR, O'Donnell E, Raje N, Yee AJ, Patterson CJ, Hunter ZR, Treon SP. Long-term follow-up of ibrutinib monotherapy in treatment-naive patients with Waldenstrom macroglobulinemia. Leukemia. 2022 Feb;36(2):532-539. doi: 10.1038/s41375-021-01417-9. Epub 2021 Sep 16. PMID 34531537
- [Background] Dimopoulos MA, Tedeschi A, Trotman J, Garcia-Sanz R, Macdonald D, Leblond V, Mahe B, Herbaux C, Tam C, Orsucci L, Palomba ML, Matous JV, Shustik C, Kastritis E, Treon SP, Li J, Salman Z, Graef T, Buske C; iNNOVATE Study Group and the European Consortium for Waldenstrom's Macroglobulinemia. Phase 3 Trial of Ibrutinib plus Rituximab in Waldenstrom's Macroglobulinemia. N Engl J Med. 2018 Jun 21;378(25):2399-2410. doi: 10.1056/NEJMoa1802917. Epub 2018 Jun 1. PMID 29856685
- [Background] Trotman J, Opat S, Gottlieb D, Simpson D, Marlton P, Cull G, Munoz J, Tedeschi A, Roberts AW, Seymour JF, Atwal SK, Yu Y, Novotny W, Holmgren E, Tan Z, Hilger JD, Huang J, Tam CS. Zanubrutinib for the treatment of patients with Waldenstrom macroglobulinemia: 3 years of follow-up. Blood. 2020 Oct 29;136(18):2027-2037. doi: 10.1182/blood.2020006449. PMID 32698195
- [Background] Kastritis E, Gavriatopoulou M, Kyrtsonis MC, Roussou M, Hadjiharissi E, Symeonidis A, Repoussis P, Michalis E, Delimpasi S, Tsatalas K, Tsirigotis P, Vassou A, Vervessou E, Katodritou E, Gika D, Terpos E, Dimopoulos MA. Dexamethasone, rituximab, and cyclophosphamide as primary treatment of Waldenstrom macroglobulinemia: final analysis of a phase 2 study. Blood. 2015 Sep 10;126(11):1392-4. doi: 10.1182/blood-2015-05-647420. No abstract available. PMID 26359434
- [Background] Treon SP, Soumerai JD, Branagan AR, Hunter ZR, Patterson CJ, Ioakimidis L, Chu L, Musto P, Baron AD, Nunnink JC, Kash JJ, Terjanian TO, Hyman PM, Nawfel EL, Sharon DJ, Munshi NC, Anderson KC. Lenalidomide and rituximab in Waldenstrom's macroglobulinemia. Clin Cancer Res. 2009 Jan 1;15(1):355-60. doi: 10.1158/1078-0432.CCR-08-0862. PMID 19118065
- [Background] Paludo J, Abeykoon JP, Shreders A, Ansell SM, Kumar S, Ailawadhi S, King RL, Koehler AB, Reeder CB, Buadi FK, Dispenzieri A, Lacy MQ, Dingli D, Witzig TE, Go RS, Gonsalves WI, Kourelis T, Warsame R, Leung N, Habermann TM, Hayman S, Lin Y, Kyle RA, Rajkumar SV, Gertz MA, Kapoor P. Bendamustine and rituximab (BR) versus dexamethasone, rituximab, and cyclophosphamide (DRC) in patients with Waldenstrom macroglobulinemia. Ann Hematol. 2018 Aug;97(8):1417-1425. doi: 10.1007/s00277-018-3311-z. Epub 2018 Apr 3. PMID 29610969
- [Background] Castillo JJ, Abeykoon JP, Gustine JN, Zanwar S, Mein K, Flynn CA, Demos MG, Guerrera ML, Kofides A, Liu X, Munshi M, Tsakmaklis N, King R, Yang G, Hunter ZR, Advani RH, Palomba ML, Ansell SM, Gertz MA, Kapoor P, Treon SP. Partial response or better at six months is prognostic of superior progression-free survival in Waldenstrom macroglobulinaemia patients treated with ibrutinib. Br J Haematol. 2021 Feb;192(3):542-550. doi: 10.1111/bjh.17225. Epub 2020 Nov 18. PMID 33207010
- [Background] 2020 EHA EP1194
- [Background] 2021 ASCO 8049